CLINICAL TRIAL: NCT00454480
Title: A Programme of Treatment Development for Older Patients With Acute Myeloid Leukemia and High Risk Myelodysplastic Syndrome
Brief Title: Combination Chemotherapy With or Without Gemtuzumab Ozogamicin or Tipifarnib in Treating Patients With Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000526121; UHW-AML16; EU-20677; ISRCTN11036523; EUDRACT-2005-002846-14; MREC-CU106
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: untreated adult acute myeloid leukemia; de novo myelodysplastic syndromes; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes; refractory anemia with excess blasts; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — Alemtuzumab; Arsenic Trioxide; Azacitidine; Busulfan; Clofarabine; Cytarabine; Daunorubicin; fludarabine phosphate; Gemtuzumab; Melphalan; tipifarnib; DNA Methylation; Cytogenetic Analysis; Gene Expression Profiling; Immunologic Techniques

INTERVENTIONS:
Biological: alemtuzumab
Drug: arsenic trioxide
Drug: azacitidine
Drug: busulfan
Drug: clofarabine
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: fludarabine phosphate
Drug: gemtuzumab ozogamicin
Drug: melphalan
Drug: tipifarnib
Genetic: DNA methylation analysis
Genetic: cytogenetic analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Other: diagnostic laboratory biomarker analysis
Other: immunologic technique
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as gemtuzumab ozogamicin, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with gemtuzumab ozogamicin or tipifarnib may kill more cancer cells.

PURPOSE: This randomized phase II/III trial is studying different combination chemotherapy regimens to compare how well they work when given with or without gemtuzumab ozogamicin or tipifarnib in treating patients with acute myeloid leukemia or high-risk myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary (patients considered fit for intensive treatment)

* Compare the efficacy and toxicity of daunorubicin hydrochloride and cytarabine (DA) vs daunorubicin hydrochloride and clofarabine (DClo) as induction therapy in older patients with acute myeloid leukemia or high-risk myelodysplastic syndromes.
* Assess the value of gemtuzumab ozogamicin when given in combination with DA or DClo during course 1 of induction therapy.
* Compare a total of two vs three courses of treatment in patients who achieve at least partial remission (< 15% blasts) after course 1 of induction therapy.
* Compare the use of demethylation maintenance therapy comprising azacitidine vs no maintenance therapy in these patients.
* Assess the value of reduced-intensity allogeneic stem cell transplantation as consolidation in patients with matched donors.

Primary (patients considered unfit for intensive treatment)

* Compare the efficacy and toxicity of low-dose cytarabine with vs without gemtuzumab ozogamicin in these patients.
* Compare the efficacy and toxicity of low-dose cytarabine with vs without arsenic trioxide in these patients.
* Compare the efficacy and toxicity of low-dose cytarabine vs low-dose clofarabine in these patients.

Secondary

* Evaluate the relevance of the presence of a cytogenetic abnormality in the bone marrow of patients in morphological remission.
* Correlate molecular detection of FLT3 and RAS mutation, genetic signature, and resistance protein status with response to treatment.
* Evaluate methods of minimal residual disease monitoring.
* Correlate gene methylation status with treatment with maintenance azacitidine.

OUTLINE: This is a randomized, controlled, factorial design, prospective, multicenter study. Patients are stratified according to age (< 60 years vs 60-64 years vs 65-69 years vs 70-74 years vs ≥ 75 years), performance status, WBC count (0-9.9,000/mm³ vs 10-49.9,000/mm³ vs 50-99.9,000/mm³ vs ≥ 100,000/mm³), and type of disease (de novo acute myeloid leukemia [AML] vs secondary AML vs high-risk myelodysplastic syndromes). Patients receive treatment according to disease status (fit for intensive treatment vs unfit for intensive treatment).

* Intensive treatment (for patients considered fit for intensive treatment):

  * Induction therapy: Patients are randomized to 1 of 4 treatment arms.

    * Arm I: For course 1, patients receive daunorubicin hydrochloride (DH) IV over 1 hour on days 1, 3, and 5 and cytarabine IV twice daily on days 1-10. For course 2, patients receive DH as in course 1 and cytarabine IV twice daily on days 1-8. Courses are 4 weeks in duration.
    * Arm II: Patients receive DH IV over 1 hour on days 1, 3, and 5 and clofarabine IV over 1 hour on days 1-5. Treatment repeats every 4 weeks for 2 courses.
    * Arm III: For course 1, patients receive DH IV over 1 hour on days 1, 3, and 5, cytarabine IV twice daily on days 1-10, and gemtuzumab ozogamicin (GO) IV over 2 hours on day 1. For course 2, patients receive DH as in course 1 and cytarabine IV twice daily on days 1-8. Courses are 4 weeks in duration.
    * Arm IV: For course 1, patients receive DH and clofarabine as in arm II and GO as in arm III. For course 2, patients receive DH and clofarabine as in arm II. Courses are 4 weeks in duration.

Patients who fail to achieve partial remission (PR) or complete remission (CR) after course 1 but achieve CR after course 2 receive a third course of chemotherapy comprising DH IV over 1 hour on days 1 and 3 and cytarabine IV twice daily on day 1-5. Patients then proceed to randomization for maintenance therapy.

Patients who achieve PR or CR after course 1 and are in CR after course 2 are randomized to receive or not receive a third course of chemotherapy (as above). Patients then proceed to randomization for maintenance therapy.

Patients who have an HLA-matched donor may proceed to nonintensive allogeneic stem cell transplantation (ASCT).

* Nonintensive ASCT: Patients receive a nonintensive allograft comprising 1 of 2 mini-allograft protocols.

  * Protocol 1: Patients receive fludarabine on days -9 to -5, busulfan on days -3 and -2, and alemtuzumab on days -5 to -1. Patients undergo ASCT on day 0.
  * Protocol 2: Patients receive fludarabine on days -7 to -3, melphalan on day -2, and alemtuzumab on days -8 to -4. Patients undergo ASCT on day 0.
* Maintenance Therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive azacitidine subcutaneously (SC) once daily on days 1-5. Treatment repeats every 6 weeks for 9 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients do not receive maintenance therapy.

    * Nonintensive treatment (for patients considered unfit for intensive treatment): Patients are randomized to 1 of 4 treatment arms.
* Arm I: Patients receive low-dose cytarabine (LDC) SC twice daily on days 1-10.
* Arm II: Patients receive LDC as in arm I and GO IV over 2 hours on day 1.
* Arm III: Patients receive low-dose clofarabine IV over 1 hour once daily on days 1-5.
* Arm IV: Patients receive LDC as in arm I and arsenic trioxide IV over 1-2 hours on days 1-5, 9, and 11.

Treatment in all arms repeats every 4-6 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Bone marrow is collected at diagnosis and examined for characterization of FLT3 and RAS mutations by immunophenotyping, gene expression by DNA microarray, and cytogenetic analysis. Blood samples are collected at baseline and after 18, 36, and 54 weeks of treatment for assessment of gene methylation status.

After completion of study therapy, patients are followed at 6 and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML) meeting the following criteria:

    * De novo or secondary AML
    * No acute promyelocytic leukemia
  * High-risk myelodysplastic syndromes (> 10% marrow blasts; refractory anemia with excess blasts-2)
  * No blast transformation of chronic myeloid leukemia
* Patients ≤ 60 years of age may be eligible provided they are considered unfit for clinical trial MRC-AMLI5

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* AST and ALT ≤ 2 times upper limit of normal (ULN) (for patients receiving gemtuzumab ozogamicin)
* Bilirubin ≤ 2 times ULN (for patients receiving gemtuzumab ozogamicin)
* Creatinine normal (for patients receiving clofarabine)
* No other concurrent active malignancy except basal cell carcinoma

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic chemotherapy for AML

  * Hydroxyurea or similar low-dose therapy to control WBC count prior to initiation of intensive therapy allowed
* No concurrent enzyme anticonvulsants, including phenytoin, phenobarbital, primidone, carbamazepine, or oxcarbazepine (for patients receiving tipifarnib)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2006-08; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Overall survival
Achievement of complete remission and reasons for failure
Duration of remission, relapse rates, and deaths
Hematological and nonhematological toxicity
Supportive care requirements (and other aspects of health economics)

CONTACTS AND LOCATIONS:
Overall Officials: Alan K. Burnett, MD, FRCP, Study Chair — University Hospital of Wales
Locations (96):
- United Kingdom (96):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Queen's Hospital, Burton-on-Trent, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St. Helier Hospital, Carshalton, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Countess of Chester Hospital, Chester, England
  - Chesterfield Royal Hospital, Chesterfield, England
  - Saint Richards Hospital, Chichester, England
  - Walsgrave Hospital, Coventry, England
  - Mayday University Hospital, Croydon, England
  - Derbyshire Royal Infirmary, Derby, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Dorset County Hospital, Dorchester, England
  - Russells Hall Hospital, Dudley, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Medway Maritime Hospital, Gillingham Kent, England
  - Harrogate District Hospital, Harrogate, England
  - Northwick Park Hospital, Harrow, England
  - Hemel Hempstead General, Hemel Hempstead, England
  - Wycombe General Hospital, High Wycombe, England
  - Hull Royal Infirmary, Hull, England
  - Ipswich Hospital, Ipswich, England
  - West Middlesex University Hospital, Isleworth, England
  - Kettering General Hosptial, Kettering, Northants, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Crosshouse Hospital, Kilmarnock, England
  - Leeds General Infirmary, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - UCL Cancer Institute, London, England
  - University Hospital Lewisham, London, England
  - Queen Elizabeth Hospital - Woolwich, London, England
  - King's College Hospital, London, England
  - St. George's Hospital, London, England
  - University College Hospital - London, London, England
  - Maidstone Hospital, Maidstone, England
  - Manchester Royal Infirmary, Manchester, England
  - Christie Hospital, Manchester, England
  - Trafford General Hospital, Manchester, England
  - Borders General Hospital, Melrose, England
  - Arrowe Park Hospital, Metropolitan Borough of Wirral, England
  - James Paget Hospital, Norfolk, England
  - Nottingham City Hospital, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Whiston Hospital, Prescot Merseyside, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Hope Hospital, Salford, England
  - Salisbury District Hospital, Salisbury, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Southport and Formby District General Hospital, Southport, England
  - Staffordshire General Hospital, Stafford, England
  - Sunderland Royal Hospital, Sunderland, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Hillingdon Hospital, Uxbridge, England
  - Sandwell General Hospital, West Bromwich, England
  - Worcester Royal Hospital, Worcester, England
  - Worthing Hospital, Worthing, England
  - Cancer Care Center, York, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Monklands General Hospital, Airdrie, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Victoria Infirmary, Glasgow, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Victoria Hospital, Kirkcaldy, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Dorset Cancer Centre, Wakefield, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - South West Wales Cancer Institute, Swansea, Wales
  - Hereford Hospitals, Hereford
  - Wexham Park Hospital, Slough, Berkshire
  - Kingston Hospital, Surrey